CLINICAL TRIAL: NCT02987400
Title: Phase II Single-arm "Window-of-opportunity" Study of a Combination of Obinutuzumab (GA-101) and Venetoclax (ABT-199) in Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Combination of Obinutuzumab and Venetoclax in Relapsed or Refractory DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_NHL-15B; 2016-001760-10 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: DLBCL; GA-101; ABT-199; relapsed DLBCL; refractory DLBCL; AGMT; Diffuse large B-cell lymphoma; window of opportunity
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Obinutuzumab is given in a 21 day cycle intravenously starting at 1000 mg on day 1, 8 and 15 in cycle 1 and on day 1 of each following cycle Venetoclax is given orally at a dose of 800mg daily from day 1 of the first cycle.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Venetoclax — 3 cycles followed by 9 cycles consolidation if not transplant eligible
  Other Names: GA-101
Drug: Obinutuzumab — 3 cycles followed by 9 cycles consolidation if not transplant eligible
  Other Names: Gazyvaro

SUMMARY:
The purpose of this study is to evaluate the clinical activity and tolerability of a combination of obinutuzumab plus venetoclax in patients with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
The study will have a 6 patient run-in phase to determine safety and to adjust treatment. Once the sixth patient has completed 21 days of treatment, withdrawn due to toxicity, or died, a formal review will be undertaken by the sponsor (AGMT). Enrolment will be halted until review is completed. If one (1) treatment related death is reported or three (3) or more patients experience CTC grade 4 events other than neutropenia, anemia, or thrombocytopenia, the study will be stopped for further recruitment. If the stopping criteria are not met, enrollment will be continued. A futility analysis will be conducted when the first 10 patients have been evaluated for response: If at least 2 patients had an objective response (CR or PR), the study will be continued.

The combination treatment will be repeated for up to 3 cycles. The first response assessment (including PET-CT) will be performed after the first cycle of obinutuzumab-venetoclax and patients with at least stable disease (SD) or better will be given another 2 cycles of therapy and then have assessment after a total of 3 cycles. Patients with complete or partial remission (CR, PR) after 3 cycles of therapy will either go on to transplant or receive 9 further cycles of the combination therapy (if transplant ineligible). Patients with progressive disease at any time-point or stable disease after 3 cycles will be taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse large B-cell lymphoma (DLBCL)

  * with histologically confirmed relapse within 12 months after having achieved a PR or CR with initial R-anthracycline containing therapy, or
  * with refractoriness to initial R-anthracycline containing therapy (not achieving at least a partial response)
  * Bcl-2 protein expression detected by immunohistochemistry.
* Adequate organ function,
* At least one bi-dimensionally measurable lesion on CT scan defined as > 1.5 cm in its longest dimension.
* Confirmed availability of archival or freshly biopsied tumor tissue meeting protocol-defined-specifications prior to study enrolment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Adequate hematologic function (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator)

Exclusion Criteria:

* Patient has received any other investigational treatment within 28 days before study entry.
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of obinutuzumab or venetoclax.
* DLBCL transformed from other malignancies or CD20 negative DLBCL.
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤ 4 weeks prior to Cycle 1 Day 1.
* Ongoing corticosteroid use > 30 mg/day of prednisone or equivalent. Patients who received corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks duration prior to randomization (Cycle 1 Day 1). Patients may have received a brief (< 7 days) course of systemic steroids (≤ 100 mg prednisone equivalent) prior to initiation of study therapy for control of lymphoma-related symptoms.
* ECOG performance status ≥ 3.
* Female patients who are pregnant or breast-feeding.
* Acute or uncontrolled chronic infections.
* Known diagnosis of HIV
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML.
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications.
* Any sensory or motor peripheral neuropathy greater than or equal to Grade 2.
* Known history of any of the following cardiovascular conditions:

  * myocardial infarction within 2 years of study entry,
  * New York Heart Association (NYHA) Class III or IV heart failure,
  * evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities,
  * recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50% .
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease.
* Patients with transformed lymphoma.
* Primary CNS lymphoma.
* Vaccination with live vaccines within 28 days prior to treatment.
* History of other malignancy that could affect compliance with the protocol or interpretation of results (Patients with a history of curatively treated basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible).
* Patients with a malignancy that has been treated with surgery alone with curative intent will also be excluded, unless the malignancy has been in documented remission without treatment for ≥ 3 years prior to enrollment.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient.
* Significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day 1.
* Requires the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin).
* Received the following agents within 7 days prior to the first dose of venetoclax:

  * CYP3A inhibitors such as fluconazole, ketoconazole, and clarithromycin
  * Strong CYP3A inducers such as rifampin, carbamazepine
* Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit within 3 days prior to the first dose of venetoclax.
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Presence of positive test results for Hepatitis B, Hepatitis C and CMV.
* Recent major surgery (within 6 weeks prior to the start of Cycle 1 Day 1), other than for diagnosis.
* Any of the following abnormal laboratory values:

  * Calculated creatinine clearance < 50 mL/min with the use of the 24-hour creatinine clearance or modified Cockcroft-Gault equation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Clinical activity and tolerability | After 3 cycles of treatment (9 weeks)
  Objective response rate (complete or partial responses; best response) defined by PET/CT scan and bone marrow examination examination after 3 cycles.

SECONDARY OUTCOMES:
Safety: Incidence of dose-limiting toxicities | 9 weeks induction plus maximum of 27 weeks consolidation
  Incidence of dose-limiting toxicities of the combination treatment.
Response duration | From first documented response until end of follow up (max 108 weeks)
Progression-free survival | 72 weeks after last patient last visit
Overall survival | 72 weeks after last patient last visit
Ability to proceed to further stem cell transplantation | After 3 cycles of treatment (9 weeks)
  Assessed by number of eligible patients reaching transplant
Genetically/biomarker defined subgroups | 72 weeks after last patient last visit
  Identification of genetically/biomarker defined subgroups regarding response and survival

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Jäger, MD, Study Director — Medical University of Vienna
Locations (6):
- Austria (6):
  - UK Graz: Universitätsklinik für Innere Medizin; Klinische Abteilung für Hämatologie, Graz
  - Medizinische Universität Innsbruck Univ.-Klinik für Innere Medizin V Hämatologie und Onkologie, Innsbruck
  - Kepler Universitätsklinikum Linz, Med Campus III.,Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz
  - Universitätsklinik für Innere Med. III, PMU Salzburg, Salzburg
  - AKH Meduni Wien Universitätsklinik für Innere Medizin I Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna
  - Klinikum Wels-Grieskirchen, Abteilung für Innere Medizin IV, Wels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.agmt.at